CLINICAL TRIAL: NCT02559401
Title: Validation of Edema-invariant Multi-shell High Angular Resolution Diffusion Imaging (msHARDI)-Based Tractography With Intra-operative Cortical Stimulation
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 42313
Record Dates: First submitted 2015-06-19; First posted 2015-09-24 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Brain Lesions
Keywords: Eloquent cortex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: MRI
Other: Neurocognitive battery

SUMMARY:
Currently, standard-of-care tractography is based on information obtained from diffusion tensor imaging (DTI). DTI is a diffusion magnetic resonance imaging (dMRI) technique that is routinely obtained on neurosurgical patients to assist in pre-operative planning. The primary objective of the proposed study is to determine the ability of msHARDI-based tractography to discern fibers in edematous brain regions.

ELIGIBILITY:
Inclusion Criteria:

* brain lesions, including but not limited to tumors, epileptic foci, and vascular abnormalities, in or around eloquent brain regions (i.e., motor, language);
* clinical need for pre-operative 'advanced imaging' (which includes conventional DTI);
* age between 18-80 years of age;
* male or female gender. Eloquent regions include: Temporal and frontal lobes (speech/language); bilateral occipital lobes (vision); bilateral parietal lobes (sensation); and bilateral motor cortex (movement).

Exclusion Criteria:

* a contraindication for obtaining an MRI scan (e.g. implanted devices, retrained foreign body)
* pregnancy
* absence of the capacity to make medical decisions or provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with brain lesions near eloquent cortex
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-06; Primary Completion 2020-10-01 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects providing completion of the neurocognitive battery | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Brem, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States